CLINICAL TRIAL: NCT02943213
Title: A Single Center, Single Dose, Open-Label, Two-Period Replicate Pilot Study to Investigate Intra-subject Variability in the Bioavailability of a Formulation Containing Chlorpromazine Hydrochloride (25 mg Sugar Coated Tablets) in at Least 16 Healthy Males and Females Under Fasting Conditions
Brief Title: Assessment of Intra-subject Variability in the Bioavailability of Chlorpromazine Hydrochloride
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cycle Pharmaceuticals Ltd. (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CT-004; PXL231486 (Other: PAREXEL (Clinical Trial Unit))
Record Dates: First submitted 2016-10-21; First posted 2016-10-24 (Estimated); Results first posted 2017-10-13 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-10

CONDITIONS: Anti-Psychotic; Management of Manifestations of Psychotic Disorders; Treatment of Schizophrenia; Control Nausea and Vomiting; Relief of Restlessness and Apprehension Before Surgery; Acute Intermittent Porphyria; Adjunct in the Treatment of Tetanus; Control Manifestations of the Manic Type of Mani-depressive Illness; Relief of Intractable Hiccups
Keywords: Chlorpromazine; Hydrochloride; Chlorpromazine Hydrochloride; Bioavailability; Variability; Variable; Absorption; USL Pharma; USL; Healthy; South Africa; Cycle; Anti-Psychotic
MeSH Terms: conditions — Vomiting; Porphyria, Acute Intermittent | interventions — Chlorpromazine; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Period 1 (Experimental): First dosing period in which all enrolled subjects are administered a single dose of 25 mg Chlorpromazine Hydrochloride Tablet.
  Interventions: Drug: Chlorpromazine Hydrochloride
- Treatment Period 2 (Experimental): Second dosing period in which all enrolled subjects are administered a single dose of 25 mg Chlorpromazine Hydrochloride Tablet.
  Interventions: Drug: Chlorpromazine Hydrochloride

INTERVENTIONS:
Drug: Chlorpromazine Hydrochloride — Chlorpromazine Hydrochloride (25 mg Tablet) - Generic US Applicant holder is USL Pharma Inc.
  Other Names: Trade name: Chlorpromazine Hydrochloride 25 mg Tablets, USP

SUMMARY:
Cycle Pharmaceuticals Ltd. (Cycle) is developing an oral tablet formulation of Chlorpromazine Hydrochloride and intends to conduct bioequivalence trials to demonstrate its similarity to the RLD.

The aim of this pilot study is to investigate intrasubject variability in the bioavailability of Chlorpromazine Hydrochloride 25 mg sugar coated tablets.

Cycle aims to demonstrate that Chlorpromazine Hydrochloride has a shallow dose response curve and a wide safety margin. This will then allow for the modification of bioequivalence acceptance criteria in future pivotal studies which will reduce the number of participants required whilst still maintaining assurance of safety and efficacy.

Pilot Subjects (n): 20 Periods: 2 (2xR) Dosing: Single-dose Strength: 25 mg Test Product: N/A Reference: USL PHARMA Chlorpromazine Hydrochloride Analytes (in plasma): Chlorpromazine; 7-Hydroxychlorpromazine Bioequivalence based on 90% CI (Cmax, AUC): Standard; 80.00 - 125.00%

DETAILED DESCRIPTION:
This will be a single-dose, open-label, two-period replicate pilot study with orally administered chlorpromazine hydrochloride 25 mg (sugar coated tablets) conducted under fasting conditions in at least 16 healthy male and female subjects at a single study center.

Up to 20 eligible subjects will be enrolled in the study with 16 evaluable subjects to complete the study.

Analytes to be measured will be Chlorpromazine and 7-hydroxy-Chlorpromazine (free) as stipulated by FDA Guidance for assessment of bioequivalence for Chlorpromazine.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females, 18 to 65 years (both inclusive) at signing of informed consent.
2. Body Mass Index (BMI) between 18.5 and 30 kg/m2 (both inclusive).
3. Body mass not less than 50 kg.
4. Medical history, vital signs, physical examination, standard 12-lead electrocardiogram (ECG) and laboratory investigations must be clinically acceptable or within laboratory reference ranges for the relevant laboratory tests, unless the investigator considers the deviation to be irrelevant for the purpose of the study.
5. Non-smokers.
6. Females, if:

   * Not of childbearing potential, e.g., has been surgically sterilized, undergone a hysterectomy, amenorrhea for ≥ 12 months and considered post-menopausal, Note: In postmenopausal women, the value of the serum pregnancy test may be slightly increased. This test will be repeated to confirm the results. If there is no increase indicative of pregnancy, the female will be included in the study.

   OR
   * Of childbearing potential, the following conditions are to be met:
   * Negative pregnancy test
   * If this test is positive, the subject will be excluded from the study. In the rare circumstance that a pregnancy is discovered after the subject received IMP, every attempt must be made to follow her to term.
   * Not lactating
   * Abstaining from sexual activity (if this is the usual lifestyle of the subject) or must agree to use an accepted method of contraception, and agree to continue with the same method throughout the study. Examples of reliable methods of contraception include non-hormonal intrauterine device, and barrier methods combined with an additional contraceptive method.

   In this study the concomitant use of hormonal contraceptives is NOT allowed. Other methods, if considered by the investigator as reliable, will be accepted.
7. Written consent given for participation in the study.

Exclusion Criteria:

1. Evidence of psychiatric disorder, antagonistic personality, poor motivation, emotional or intellectual problems likely to limit the validity of consent to participate in the study or limit the ability to comply with protocol requirements.
2. Current alcohol use > 21 units of alcohol per week for males and > 14 units of alcohol per week for females.
3. Consumption of more than 5 cups of coffee (or equivalent amounts of caffeine) per day.
4. Regular exposure to substances of abuse (other than alcohol) within the past year.
5. Use of any medication, prescribed or over-the-counter or herbal remedies, within 2 weeks before the first administration of IMP except if this will not affect the outcome of the study in the opinion of the investigator.

   In this study the concomitant use of hormonal contraceptives is NOT allowed.
6. Participation in another study with an experimental drug, where the last administration of the previous IMP was within 8 weeks (or within 10 elimination half-lives for chemical entities or 2 elimination half-lives for antibodies or insulin), whichever is the longer) before administration of IMP in this study, at the discretion of the investigator.
7. Treatment within the previous 3 months before the first administration of IMP with any drug with a well-defined potential for adversely affecting a major organ or system.
8. A major illness during the 3 months before commencement of the screening period.
9. History of hypersensitivity or allergy to the IMP or its excipients or any related medication including phenothiazines or other anti-psychotics or anti-emetics.
10. History of extrapyramidal symptoms.
11. History of liver or renal dysfunction, epilepsy, Parkinson's disease, hypothyroidism, cardiac failure, phaeochromocytoma, myasthenia gravis, prostate hypertrophy.
12. Familial history of deep vein thrombosis.
13. Hereditary problems of galactose intolerance, Lapp lactase deficiency.
14. History of QT prolongation or signs of QT prolongation on ECG.
15. History of bronchial asthma or any other bronchospastic disease.
16. History of convulsions.
17. History of porphyria.
18. Relevant history or laboratory or clinical findings indicative of acute or chronic disease, likely to influence study outcome.
19. Donation or loss of blood equal to or exceeding 500 mL during the 8 weeks before the first administration of IMP.
20. Diagnosis of hypotension made during the screening period.
21. Diagnosis of hypertension made during the screening period or current diagnosis of hypertension.
22. Resting pulse of > 100 beats per minute or < 40 beats per minute during the screening period, either supine or standing.
23. Positive testing for HIV and Hepatitis B and Hepatitis C.
24. Positive urine screen for drugs of abuse. In case of a positive result the urine screen for drugs of abuse may be repeated once at the discretion of the investigator.
25. Positive urine screen for tobacco use.
26. Female subjects that are pregnant (positive pregnancy test) or breastfeeding.
27. Difficulty in swallowing.
28. Any specific investigational product safety concern.
29. Vulnerable subjects, e.g., persons in detention.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-11; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Yolandi Swart, FCPHM(SA), Principal Investigator — Bloemfontein Early Phase Clinical Unit, PAREXEL International (South Africa)
Locations (1):
- Farmovs Parexel, Bloemfontein, Kampuslaan Suid, South Africa

IPD SHARING:
Plan to Share IPD: No
participants are healthy volunteers.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study volunteers each received a single dose of 25 mg Chlorpromazine Hydrochloride Tablet in both treatment periods.
Groups:
- Chlorpromazine 25 mg: All enrolled subjects are administered a single dose of 25 mg Chlorpromazine Hydrochloride Tablet.
  Chlorpromazine Hydrochloride: Chlorpromazine Hydrochloride (25 mg Tablet) - Generic US Applicant holder is USL Pharma Inc.
Period: Treatment Period 1
Arm/Group | Chlorpromazine 25 mg
Started | 20
Completed | 20
Not Completed | 0
Period: Treatment Period 2
Arm/Group | Chlorpromazine 25 mg
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Chlorpromazine 25 mg
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 4
  Black | 16
Region of Enrollment [Count of Participants; unit: Participants]
  South Africa | 20

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) - Chlorpromazine
Description: Time Frame = sampling times.
Time Frame: 0, 0.5, 1, 1.3, 1.6, 2, 2.5, 3, 4, 5, 6, 9, 12, 16, 24, 36, 48, 72 and 96 hours
Population: All subjects who completed the PK blood sampling for this study and for whom primary PK parameters were calculated for both treatment periods were included in the statistical PK analysis of the study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Groups:
- Treatment Period 1; Treatment Period 2: All enrolled subjects are administered a single dose of 25 mg Chlorpromazine Hydrochloride Tablet.
  Chlorpromazine Hydrochloride: Chlorpromazine Hydrochloride (25 mg Tablet) - Generic US Applicant holder is USL Pharma Inc.
Arm/Group | Treatment Period 1 | Treatment Period 2
Number analyzed (Participants) | 20 | 20
pg/mL | 2671 (94.5) | 2720 (69.6)

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) - 7-Hydroxy-Chlorpromazine
Description: Time Frame = sampling times.
Time Frame: 0, 0.5, 1, 1.3, 1.6, 2, 2.5, 3, 4, 5, 6, 9, 12, 16, 24, 36, 48, 72 and 96 hours
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Treatment Period 1 | Treatment Period 2
Number analyzed (Participants) | 20 | 20
pg/mL | 1539 (57.6) | 1583 (48.9)

3. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve, From Time Zero to t, Where t is the Time of the Last Quantifiable Concentration (AUC(0-t)) - Chlorpromazine
Description: Time Frame = sampling times.
Time Frame: 0, 0.5, 1, 1.3, 1.6, 2, 2.5, 3, 4, 5, 6, 9, 12, 16, 24, 36, 48, 72 and 96 hours
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | Treatment Period 1 | Treatment Period 2
Number analyzed (Participants) | 20 | 20
h*pg/mL | 18670 (91.9) | 18470 (98.0)

4. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve, From Time Zero to t, Where t is the Time of the Last Quantifiable Concentration (AUC(0-t)) - 7-Hydroxy-Chlorpromazine
Description: Time Frame = sampling times.
Time Frame: 0, 0.5, 1, 1.3, 1.6, 2, 2.5, 3, 4, 5, 6, 9, 12, 16, 24, 36, 48, 72 and 96 hours
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | Treatment Period 1 | Treatment Period 2
Number analyzed (Participants) | 20 | 20
h*pg/mL | 13280 (58.4) | 13190 (61.6)

5. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve, With Extrapolation to Infinity (AUC(0-∞)) - Chlorpromazine
Description: Time Frame = sampling times.
Time Frame: 0, 0.5, 1, 1.3, 1.6, 2, 2.5, 3, 4, 5, 6, 9, 12, 16, 24, 36, 48, 72 and 96 hours
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | Treatment Period 1 | Treatment Period 2
Number analyzed (Participants) | 20 | 20
h*pg/mL | 15790 (74.9) | 19650 (106.2)

6. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve, With Extrapolation to Infinity (AUC(0-∞)) - 7-Hydroxy-Chlorpromazine
Description: Time Frame = sampling times.
Time Frame: 0, 0.5, 1, 1.3, 1.6, 2, 2.5, 3, 4, 5, 6, 9, 12, 16, 24, 36, 48, 72 and 96 hours
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | Treatment Period 1 | Treatment Period 2
Number analyzed (Participants) | 20 | 20
h*pg/mL | 14460 (55.2) | 13740 (60.7)

7. Secondary Outcome: Time to Maximum Observed Plasma Concentration (Tmax) - Chlorpromazine
Description: Time Frame = sampling times
Time Frame: 0, 0.5, 1, 1.3, 1.6, 2, 2.5, 3, 4, 5, 6, 9, 12, 16, 24, 36, 48, 72 and 96 hours
Population: as for outcome 1
Measure: Median (Full Range); unit: hr
Arm/Group | Treatment Period 1 | Treatment Period 2
Number analyzed (Participants) | 20 | 20
hr | 1.33 [1 to 2] | 1.33 [1 to 5]

8. Secondary Outcome: Time to Maximum Observed Plasma Concentration (Tmax) - 7-Hydroxy-Chlorpromazine
Description: Time Frame = sampling times
Time Frame: 0, 0.5, 1, 1.3, 1.6, 2, 2.5, 3, 4, 5, 6, 9, 12, 16, 24, 36, 48, 72 and 96 hours
Population: as for outcome 1
Measure: Median (Full Range); unit: hr
Arm/Group | Treatment Period 1 | Treatment Period 2
Number analyzed (Participants) | 20 | 20
hr | 2.00 [1.33 to 3.00] | 1.83 [1.00 to 3.00]

9. Secondary Outcome: Terminal Elimination Rate Constant (λz) - Chlorpromazine
Description: Time Frame = sampling times
Time Frame: 0, 0.5, 1, 1.3, 1.6, 2, 2.5, 3, 4, 5, 6, 9, 12, 16, 24, 36, 48, 72 and 96 hours
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hr
Arm/Group | Treatment Period 1 | Treatment Period 2
Number analyzed (Participants) | 20 | 20
1/hr | 0.05060 (17.9) | 0.04117 (32.6)

10. Secondary Outcome: Terminal Elimination Rate Constant (λz) - 7-Hydroxy-Chlorpromazine
Description: Time Frame = sampling times
Time Frame: 0, 0.5, 1, 1.3, 1.6, 2, 2.5, 3, 4, 5, 6, 9, 12, 16, 24, 36, 48, 72 and 96 hours
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hr
Arm/Group | Treatment Period 1 | Treatment Period 2
Number analyzed (Participants) | 20 | 20
1/hr | 0.07153 (19.5) | 0.07025 (19.8)

11. Secondary Outcome: Apparent Terminal Elimination Half-life (t1/2) - Chlorpromazine
Description: Time Frame = sampling times
Time Frame: 0, 0.5, 1, 1.3, 1.6, 2, 2.5, 3, 4, 5, 6, 9, 12, 16, 24, 36, 48, 72 and 96 hours
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Treatment Period 1 | Treatment Period 2
Number analyzed (Participants) | 20 | 20
hr | 13.70 (17.7) | 16.84 (40.7)

12. Secondary Outcome: Apparent Terminal Elimination Half-life (t1/2) - 7-Hydroxy-Chlorpromazine
Description: Time Frame = sampling times
Time Frame: 0, 0.5, 1, 1.3, 1.6, 2, 2.5, 3, 4, 5, 6, 9, 12, 16, 24, 36, 48, 72 and 96 hours
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Treatment Period 1 | Treatment Period 2
Number analyzed (Participants) | 20 | 20
hr | 9.690 (31.8) | 9.867 (28.1)

ADVERSE EVENTS:
Time Frame: From first visit first dose until post-study visit.
Arm/Group | Treatment Period 1 | Treatment Period 2
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 2/20 | 1/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Period 1 (N=20) | Treatment Period 2 (N=20)
Arthralgia Left Index Finger (Musculoskeletal and connective tissue disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Soft Tissue Injury Right Side of Body (Injury, poisoning and procedural complications) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No